CLINICAL TRIAL: NCT01804335
Title: Exploratory Study to Evaluate the Safety and Efficacy of CD5789 in Subjects With Early Stage Cutaneous T-Cell Lymphoma
Brief Title: CD5789 in Early Cutaneous T-Cell Lymphoma (CTCL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0710; NCI-2014-01377 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-03-01; First posted 2013-03-05 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Lymphoma
Keywords: Lymphoma; Early Stage Cutaneous T-Cell Lymphoma; CTCL; CD5789 0.01% cream
MeSH Terms: conditions — Lymphoma | interventions — trifarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CD5789 0.01% Cream (Experimental): CD5789 0.01% cream applied on the lesions once daily for twelve weeks.
  Interventions: Drug: CD5789 0.01% Cream

INTERVENTIONS:
Drug: CD5789 0.01% Cream — CD5789 0.01% cream applied on the lesions once daily for twelve weeks.

SUMMARY:
The goal of this clinical research study is to learn if CD5789 is safe and tolerable when given to patients with early stage CTCL.

CD5789 is designed to attach to tumor cells and change their genetic material. This may stop the growth of the tumor cells.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will apply CD5789 cream 1 time each day. You should do this after you wash the area.

During your first study visit, the study staff will select which lesions you will apply cream to. The study staff will tell you how much cream to apply.

On Day 1, the study staff will apply the study drug on half of the lesions. You will apply the study drug to the rest of the lesions while the study staff watches. In a diary, the study staff will write down the time you applied the study drug. You must write down this information in the diary when you apply the study drug at home. On your Week 1 visit, you will apply the study drug at the clinic while the study staff watches.

You will use gloves to apply the study drug in a thin film on the lesions. Be careful not to overlap healthy skin. You should massage the study drug gently into the skin. If someone helps you apply the study drug, they must also wear gloves.

Bring the diary with you to each visit. You should return all unused study drug and/or empty tubes at each study visit.

You must avoid exposing the treated areas to the sun (you should wear clothing to cover these areas). You should also not swim or take a bath while on study, but you can take a shower at least 2 hours after you apply the drug.

If your skin is dry, you will be given a moisturizer (such as Cetaphil Restoraderm Skin Restoring Moisturizer) to use.

Study Visits:

At all study visits, you will asked about any drugs you may be taking or any side effects you may have had.

On Day 1:

* Any skin lesions will be measured and photographed. Your private areas will be covered as much as possible, and a picture of your face will not be taken.
* You will have a skin biopsy to check the status of the disease. To perform a skin biopsy, an area will be numbed with anesthetic and a small amount of skin will be removed with a small knife. The skin biopsy will be done before you apply the study drug.
* You will have tape stripping to measure any inflammatory markers on the skin. Inflammatory markers may be related to the status of the disease. To have tape stripping, small special pieces of tape will be applied to 1 skin lesion and to an area of normal skin next to it. When the tape loses it stickiness it will be collected by the study staff.
* You will have an EKG to check your heart function.
* You will be asked about how much you itch and if you have any burning or stinging sensations after applying the study drug.
* If you can become pregnant, urine will be collected for a urine pregnancy test.

At Weeks 1, 2, 4, and 8:

* Any skin lesions will be measured and photographed.
* You will be asked about how much you itch and if you have any burning or stinging sensations after applying the study drug.

At Weeks 4 and 8, if you can become pregnant, urine will be collected for a urine pregnancy test.

Length of Study:

You may continue using the study drug for up to 12 weeks, as long as the study doctor thinks it is in your best interest. You will no longer be able to use the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over when you have completed the end-of-study visit.

All samples collected during the study will be destroyed after the study has been completed and all patients are off study.

End-of-Study Visit:

On the last day you apply the study drug (Week 12), you will have an end-of-study visit:

* You will be asked about any other drugs and treatments you may be receiving.
* You will have a physical exam, including measurement of your vital signs.
* Any skin lesions will be examined and photographed.
* Blood (about 2½ teaspoons) will be drawn for routine tests. and to tests for HIV and/or hepatitis.
* Blood (about 1 teaspoon each time) will be drawn for pharmacokinetic (PK) testing 12 hours after the study drug is applied at home PK testing measures the amount of study drug in the body at different time points.
* You will have an EKG to check your heart function.
* You will have a skin biopsy to check the status of the disease.
* You will have tape stripping to measure any inflammatory markers on the skin.
* If you can become pregnant, urine will be collected for a pregnancy test.

This is an investigational study. CD5789 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 10 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. The Subject is a male or female, who is at least 18 years of age at Screening visit.
2. The Subject has a clinical diagnosis of stable CTCL early stage (IA-IIA). The subject has :a) A known stable TNMB stage (cancer classification based on analysis of Tumors, Nodes, Metastasis and Blood), or b) Stable patch or plaque lesions that have not responded to topical treatment with corticosteroids or nitrogen mustard or which have relapsed after prior therapy.
3. The Subject presents at least 3 distinct lesions (one selected as index lesion, one dedicated to biopsy and another one dedicated to tape-stripping).
4. If the Subject is a female of childbearing potential, she agrees to use a highly contraceptive method for the duration of the study and for one month after the last product application. A highly effective method of contraception is defined by: 1) Bilateral tubal ligation 2) Combined oral contraceptives (estrogen and progesterone) implanted or injectable contraceptives, on a stable dose for at least 1 month prior to screening visit, 3) Hormonal intra-uterine device (IUD), inserted at least one month prior to the Screening visit.
5. If the Subject is female of childbearing potential, she has at Screening (at least 14 days before Baseline) and at Baseline a negative result for urine pregnancy test (UPT)having a sensitivity down to at least 25 Ul/ml for human chorionic gonadotrophin (hCG).
6. If the Subject is a female of non-childbearing potential, she has to be postmenopausal (absence of menstrual bleeding for at least one year and without any other medical reason), or presenting with a hysterectomy or a bilateral ovariectomy.
7. The Subject is willing and able to comply with all of the time commitments and procedural requirements of the clinical trial protocol.
8. The Subject has understood and signed an Informed Consent Form (ICF) at Screening, prior to an investigational procedures being performed.
9. The Subject is apprised of the Health Insurance Portability and Accountability Act (HIPAA), and is willing to share personal information and data, as verified by signing a written authorization at the screening.

Exclusion Criteria:

1. The subject has any uncontrolled or serious disease (other than CTCL), or any medical or surgical condition, that may either interfere with the interpretation of the clinical trial results, and/or put the subject at significant risk (according to Investigator's judgment) if he/she participates in the clinical trial.
2. The subject has known or suspected allergies or sensitivities to any components of the study drug (see Investigator's Brochure).
3. The subject, if female, has a positive urinary pregnancy test, is breast-feeding or is planning a pregnancy during the course of the study.
4. If the subject needs a relative to apply the study product, the relative is a female who is pregnant, lactating or intends to conceive during the clinical study or within 1 month after the last product application.
5. The subject is in an exclusion period from a previous clinical study, takes part into any other clinical trial of a drug or device, OR participated within 1 month prior to baseline.
6. The subject has used any of the following treatments or procedure before the first study treatment application (Baseline) within the wash-out periods defined below: corticoids or Aldera (imiquimod) 4 weeks; retinoids, nitrogen mustard (mechlorethamine), Carmustine (BCNU), or phototherapies 2 weeks, any systemic treatment dedicated to CTCL within 4 weeks.
7. The subject is unwilling to refrain from use of prohibited medication during the clinical trial.
8. The subject has an abnormal ECG judged clinically significant by the investigator and/or PR interval outside the range of 120 ms to 220 ms, QRS>120 ms, and corrected QT interval (QTc)>450 ms.
9. The subject presents seropositivity for hepatitis B surface antigen(HBsAG), hepatitis C virus (HCV) antibody and /or human immunodeficiency virus (HIV) 1 and 2 antibody.
10. The subject is vulnerable (such as deprived of freedom) as defined in Section 1.61 of International Conference on Harmonisation (ICH) Guideline for Good Clinical Practice (GCP).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2013-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Tolerance Score of CD5789 0.01% Cream | 12 weeks
  Data analysis based on local tolerability score evaluated at each visit with a worst tolerance score for the subject calculated at each visit. Worst tolerance score is worst score of local tolerability of all index lesions for each subject at each visit. Worst tolerance score (max local tolerance score) summarized in frequency tables to follow the evolution of this score across visits for each subject.
  Index lesion(s) evaluated at each visit for local tolerance (using a 5-point scale) from Week 1 visit to Week 12/ Early Termination visit for each index lesion. Tolerance 5-point scale from 0-No reaction to 4-Severe where the higher number the worse reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Duvic, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center — http://www.mdanderson.org